CLINICAL TRIAL: NCT02222220
Title: Metoclopramide as Treatment of Clozapine-induced Hypersalivation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, Prof. Vladimir Lerner, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLAK-14
Record Dates: First submitted 2014-08-17; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2012-01

CONDITIONS: Clozapine-induced Hypersalivation
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoclopramide (Placebo Comparator): 61 participating subjects were randomized into 2 groups: 30 received metoclopramide up to 30 mg/day and 31 received placebo, each for 4 weeks in a double-blind mode
  Interventions: Drug: Metoclopramide; Drug: placebo
- metocliopramide (Experimental): 61 participating subjects were randomized into 2 groups: 30 received metoclopramide up to 30 mg/day and 31 received placebo, each for 4 weeks in a double-blind mode
  Interventions: Drug: Metoclopramide; Drug: placebo

INTERVENTIONS:
Drug: Metoclopramide — 30 mg/day during 4 weeks
Drug: placebo

SUMMARY:
Hypersalivation (sialorrhea or ptyalism) is known as a frequent, disturbing, uncomfortable adverse effect of clozapine therapy that can lead to noncompliance. Until now there is no effective enough treatment for this side effect.

Previous studies demonstrated that different medications from the substitute benzamide derivatives group: amisulpride, sulpiride (higher selective binding to the D2/D3 dopamine receptor) and moclobemide (reversible inhibitor of monoamine oxidase A, which inhibits the deamination of serotonin, norepinephrine and dopamine) may be effective as a treatment of clozapine-induced hypersalivation (CIH). Moreover, there is another substitute benzamide derivative: metoclopramide (dopamine D2 antagonist, usually used as antiemetic medication in general medicine). The investigators hypothesis assumes that anti-salivation effect characterizes the whole group of benzamide.

The aim of this study was to examine the efficacy of metoclopramide as an optional possibility for management of CIH.

DETAILED DESCRIPTION:
Hypersalivation (sialorrhea or ptyalism) is known as a frequent, disturbing, uncomfortable adverse effect of clozapine therapy that may persist for several years. This side effect is usually dose-related. It may occur all over the day, but it is most pronounced during night sleep, since swallowing reflex is diminished, and patients usually complain of wakening with a wet pillow (sometimes called as "wet pillow" sign).

Salivation is regulated by sympathetic (adrenergic) and parasympathetic (cholinergic) tones. The phenomenon of clozapine-induced hypersalivation (CIH) remains mysterious since the drug has potent α2 antagonistic, M4 - muscarinic agonistic, and anticholinergic (M1, M2, M3, and M5) activities and each of these has a different effect on the control of salivation. While α2 antagonistic and M4 - muscarinic agonistic effects increase salivation, the anticholinergic effect leads to diminished saliva secretion. It has been reported that CIH is observed from 10 to 80% of patients according to various sources, an average rate is 30% of clozapine-treated patients. Further to the social embarrassment related to hypersalivation, additional consequences of CIH include painful parotid gland swelling and parotid duct obstruction due to the formation of calculi.

Clozapine is a second generation neuroleptic agent whose structure consists of a dibenzodiazepine derivative with a piperazinyl side chain. It has a unique neuropharmacologic profile, which is attributed to atypical antipsychotic agents with proven efficacy in refractory schizophrenia, but its widespread use is limited by adverse effects such as agranulocytosis, seizures, sedation, weight gain, and sialorrhea. Clozapine has a weak binding affinity for dopamine D1 and D2 receptors by its slightly greater preference for D1 receptors, as noted with a D1:D2 receptor binding ratio of 1:3. Furthermore the drug has potent binding affinity for serotonin receptors 5-HT1A and 5-HT2, and also antihistaminic, anticholinergic, and alpha-adrenergic antagonistic properties.

Sialorrhea is troublesome its stigmatizing nature results for a schizophrenia patient led to massive compliance problems. For management of this distressing side effect have been recommended different pharmacological agents such as α2 - adrenoreceptor agonists, including clonidine, and lofexidine, but these treatments have unwanted side effects, no proved effectiveness. They are not been routinely used. These publications show that CIH probably might have a different neurobiological basis rather than the proposed mediation by the M4 - muscarinic receptor.

Previous studies found that substitute benzamide derivatives with higher selective binding to the D2/D3 dopamine receptors - amisulpride, sulpiride as well moclobemide (reversible inhibitor of monoamine oxidase A, which inhibits the deamination of serotonin, norepinephrine and dopamine) may be effective in treatment of CIH without additional adverse effects. Unfortunately, these medications are not effective in all patients who suffered from CIH.

Metoclopramide was first described by Dr. Louis Justin-Besançon and C. Laville in 1964. It is a dopamine D2 receptor antagonist, and a mixed 5-HT3 receptor antagonist. Moreover, it is a 5-HT4 receptor agonist.

Metoclopramide is fairly often used in general medicine as an antiemetic agent. In 1979, FDA approved it for treatment of nausea and vomiting. This drug also belongs to substitute benzamide derivatives group. It is assumed that the anti-emetic activity is caused by its D2 receptor antagonism in the chemoreceptor trigger zone in the central nervous system. Dry mouth is one of its side effects. The investigators hypothesized that antisalivation effect characterizes the whole group of benzamides, and will be demonstrated also in none psychotropic agent like metoclopramide.

The aim of our study was to examine efficacy of metoclopramide as an additional agent for management of CIH and to approve our hypothesis.

Subjects and Methods The study was conducted from January 2012 to May 2014 in two large state referral institutions: Tirat Carmel Mental Health Center and the Be'er-Sheva Mental Health Center. The investigators screened 68 patients (males and females, 19-60 years old) suffering from schizophrenia and schizoaffective disorders, treated with clozapine, and suffering from hypersalivation. Of all screened subjects, 7 patients refused to take part in the study.

Inclusion criteria were: a) males and females in age 18-60 years old; b) met Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision, criteria for schizophrenia or schizoaffective disorder; c) Clozapine treatment for a minimum of 2 months; d) Constant dose of clozapine and other concomitant medications during previous 2 weeks; e) At least 2 points on the Nocturnal Hypersalivation Rating Scale (NHRS);3 f) Ability and willingness to sign informed consent for participation in the study.

Study exclusion criteria included: a) the Presence of concurrent medical conditions contributing to hypersalivation (eg, idiopathic Parkinson's disease, cerebral palsy); b) Evidence of mental retardation; c) Alcohol or drug abuse. Patients who had been treated with anticholinergic agents and continued to experience CIH were allowed to participate in the study, provided they continued to suffer from CIH of at least moderate severity. Complete medical and neurological examinations, including laboratory tests, were performed. Prior to study entry, all subjects who met the inclusion criteria provided written informed consent after receiving a full explanation regarding the nature of the study and potential risks and benefits. The study was approved by both the Tirat Carmel Mental Health Center and the Be'er Sheva Mental Health Center Institutional Review Boards.

Study Design The study was conducted in two mental health centers. In order to examine our hypothesis, the investigators used an add-on design. Sixty-one patients with schizophrenia and schizoaffective disorder (males and females, 19-60 years old), according to the DSM-IV criteria, treated with clozapine and suffering from hypersalivation, enrolled into the study (30 patients in metoclopramide group and 31 in the placebo group).

Procedure and drug administration In order to find a minimal effective dose, all subjects suffering from CIH (score >2 on Nocturnal Hypersalivation Rating Scale - NHRS) in a double blind randomized mode were treated during a week with 10 mg/day of metoclopramide or placebo. The patients without improvement continuing the study with 20 mg/day of metoclopramide or placebo during the next week. Those patients, who did not respond to this dose, were continued with 30 mg/day of metoclopramide or placebo for another week.

Hypersalivation will be assessed by subjective and objective tools. Clinical global impression (CGI) patient's self-assessment will be taken as a subjective tool while NHRS and Drooling Severity Scale (DSS) as an objective one. NHRS consists of the 5-points: 0-absent; 1-minimal (signs of saliva on the pillow in the morning); 2-mild (hypersalivation wakes the patient once during the night); 3-moderate (hypersalivation wakes the patient twice during the night), and 4-severe (hypersalivation wakes the patient at least 3 times during the night). DSS also consists of the 5-points: 1- never drools, 2 -mild, only wet lips, 3-moderate, wet on lips and chin, 4-severe, clothing becomes wet and 5 - profuse, clothing, hands, tray, and objects become wet. Assessment was performed on baseline (entering into the study) and every morning during the study period and two weeks after ceasing the add-on medications.

Clinically significant improvement was defined as a reduction of at least 30% from baseline to week 2 on the NHRS and DSS.

Participants Thirty patients from Be'er Sheva Mental Health Center and 31 from Tirat Carmel Mental Health Center have participated in the study.

The study was approved by the local Institutional Ethics Review Board ("Helsinki Committee"). Only subjects who will and able to sign a written informed consent form for participation in the study, were recruited. Confidentially was ensured by means of a number coding system, and all completed research forms were stored in a secure area.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, male or female
* DSM-IV criteria for schizophrenia
* Clozapine treatment
* At least score >2 on the Nocturnal Hypersalivation Rating Scale (NHRS)

Exclusion Criteria:

* Evidence of organic brain damage, mental retardation, alcohol or drug abuse
* Patients suffering from pheochromocytoma
* Patients suffering from Parkinson's disease

Ages: 19 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Nocturnal Hypersalivation Rating Scale (NHRS) | every week, up to 4 weeks

SECONDARY OUTCOMES:
Drooling Severity Scale (DSS) | every week, up to 4 weeks

OTHER OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | every week, up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Be'er Sheva Mental Health Center,, Beersheba, Israel

REFERENCES:
- [Background] Safferman A, Lieberman JA, Kane JM, Szymanski S, Kinon B. Update on the clinical efficacy and side effects of clozapine. Schizophr Bull 1991;17:247-261. Kaplan & Sadock's Comprehensive Textbook of Psychiatry. Philadelphia: Lippincot Williams & Wilkins, 2005. Baldessarini RJ, Huston-Lyons D, Campbell A, Marsh E, Cohen BM. Do central antiadrenergic actions contribute to the atypical properties of clozapine? Br J Psychiatry Suppl 1992:12-16. Kreinin A, Epshtein S, Sheinkman A, Tell E. Sulpiride addition for the treatment of clozapine-induced hypersalivation: preliminary study. Isr J Psychiatry Relat Sci 2005;42:61-63. Kreinin A, Novitski D, Weizman A. Amisulpride treatment of clozapine-induced hypersalivation in schizophrenia patients: a randomized, double-blind, placebo-controlled cross-over study. Int Clin Psychopharmacol 2006;21:99-103. Kreinin A, Miodownik C, Libov I, Shestakova D, Lerner V. Moclobemide treatment of clozapine-induced hypersalivation: pilot open study. Clin Neuropharmacol 2009;32:151-153. Justin-Besancon L, Laville C. [Antiemetic Action of Metoclopramide with Respect to Apomorphine and Hydergine]. C R Seances Soc Biol Fil 1964;158:723-727. Rang HP, Dale MM, Ritter JM, Moore PK. Pharmacology. 5th ed. Edinburgh: Churchill Livingstone; 2003. Sweetman S, editor. Martindale: The complete drug reference. 34th ed. London: Pharmaceutical Press; 2004. Tonini M, Candura SM, Messori E, Rizzi CA. Therapeutic potential of drugs with mixed 5-HT4 agonist/5-HT3 antagonist action in the control of emesis. Pharmacol Res 1995;31:257-260. Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull 1987;13:261-276. Chouinard G, Ross-Chouinard A, Annable L, Jones B. Extrapyramidal Symptom Rating Scale. Can J Neurol Sci (abstract) 1980;7:233.
- [Derived] Kreinin A, Miodownik C, Mirkin V, Gaiduk Y, Yankovsky Y, Bersudsky Y, Lerner PP, Bergman J, Lerner V. Double-Blind, Randomized, Placebo-Controlled Trial of Metoclopramide for Hypersalivation Associated With Clozapine. J Clin Psychopharmacol. 2016 Jun;36(3):200-5. doi: 10.1097/JCP.0000000000000493. PMID 27028980